CLINICAL TRIAL: NCT02340728
Title: A Randomized Trial of Endoscopic Biliary Co-axial Stent Placement Plus/Minus Use of Radiofrequency Ablation (RFA) for Clearance of Occluded Self Expandable Metal Stents (SEMS) in Patients With Distal Biliary Obstruction From Unresectable Biliary-pancreatic Malignancies
Brief Title: Endoscopic Biliary Co-axial Stent Placement Plus/Minus Use of Radiofrequency Ablation (RFA) for Clearance of Occluded Self Expandable Metal Stents (SEMS) in Patients With Distal Biliary Obstruction From Unresectable Biliary-pancreatic Malignancies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-260
Record Dates: First submitted 2015-01-08; First posted 2015-01-19 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2019-12

CONDITIONS: Pancreatic Cancer; Unresectable Biliary-pancreatic Malignancies
Keywords: Stent Placement; Biliary Obstruction; 14-260
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cholangiopancreatography, Endoscopic Retrograde; Radiofrequency Ablation; Self Expandable Metallic Stents

ARMS (2):
- ERCP with SEMS plus radiofrequency ablation (Experimental): Endoscopic retrograde cholangiopancreatogram (ERCP) is performed under standard conditions with cannulation of the bile duct, and demonstration on a cholangiogram the location, diameter and length of the biliary stricture. The HabibTM EndoHBP probe (EMcision, London, United Kingdom) is advanced through the working channel of a side viewing endoscope over a 0.035in guidewire, and positioned across the occluded SEMS under fluoroscopy. 7-10W are usually delivered for 90 seconds with a standard high frequency generator, followed by a 1 minute resting period. Sequential applications of RFA are applied along the entire length of the stricture with an overlap of 1cm.
  Interventions: Device: ERCP with SEMS plus radiofrequency ablation
- ERCP with SEMS alone (standard of care) (Active Comparator): Endoscopic retrograde cholangiopancreatogram (ERCP) is performed under standard conditions with cannulation of the bile duct, and demonstration on a cholangiogram the location, diameter and length of the biliary stricture. The HabibTM EndoHBP probe (EMcision, London, United Kingdom) is advanced through the working channel of a side viewing endoscope over a 0.035in guidewire, and positioned across the occluded SEMS under fluoroscopy. 7-10W are usually delivered for 90 seconds with a standard high frequency generator, followed by a 1 minute resting period.
  Interventions: Device: ERCP with SEMS alone (standard of care)

INTERVENTIONS:
Device: ERCP with SEMS plus radiofrequency ablation
  Other Names: self expandable metal stents; co-axial stent placement
  Arms: ERCP with SEMS plus radiofrequency ablation
Device: ERCP with SEMS alone (standard of care)
  Other Names: self expandable metal stents; co-axial stent placement
  Arms: ERCP with SEMS alone (standard of care)

SUMMARY:
The purpose of this study is to compare the effects good and/or bad of combining radiofrequency ablation with placement of a second stent, versus a second stent alone. The investigators will also look at the safety of the combination treatment, and see which treatment is better. In either case, the second stent will be placed inside the existing stent as is done in standard practice when treating a blocked stent for the first time.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any tumor obstructing the distal bile duct and causing an indwelling biliary SEMS
* Patients with jaundice or clinical cholangitis, with new elevation of alkaline phosphatase, total bilirubin, and imaging findings supportive of stent occlusion (loss of stent patency, debris within stent, loss of or excessive pneumobilia)
* Age ≥ 18 years

Exclusion Criteria:

* Have altered gastro-duodenal or hepatobiliary anatomy such that ERCP is felt to be unacceptably technically difficult or unsafe
* Have additional sites of biliary strictures (intrahepatic/hilar) such that ERCP stenting is felt to be unlikely to provide adequate clinical benefit
* Have cardiac pacemakers
* Have Child B/C cirrhosis
* Are pregnant
* Are unsuitable for endoscopy (either because of hemodynamic instability, respiratory distress or unsafe hematological parameters such as refractory anemia <7g/dL, thrombocytopenia <50K/mcL, or coagulopathy with INR >2.0)
* Have biliary strictures not technically amenable to endoscopic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Schattner, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- ERCP With SEMS Plus Radiofrequency Ablation: Endoscopic retrograde cholangiopancreatogram (ERCP) is performed under standard conditions with cannulation of the bile duct, and demonstration on a cholangiogram the location, diameter and length of the biliary stricture. The HabibTM EndoHBP probe (EMcision, London, United Kingdom) is advanced through the working channel of a side viewing endoscope over a 0.035in guidewire, and positioned across the occluded SEMS under fluoroscopy. 7-10W are usually delivered for 90 seconds with a standard high frequency generator, followed by a 1 minute resting period. Sequential applications of RFA are applied along the entire length of the stricture with an overlap of 1cm.
  ERCP with SEMS plus radiofrequency ablation
- ERCP With SEMS Alone (Standard of Care): Endoscopic retrograde cholangiopancreatogram (ERCP) is performed under standard conditions with cannulation of the bile duct, and demonstration on a cholangiogram the location, diameter and length of the biliary stricture. The HabibTM EndoHBP probe (EMcision, London, United Kingdom) is advanced through the working channel of a side viewing endoscope over a 0.035in guidewire, and positioned across the occluded SEMS under fluoroscopy. 7-10W are usually delivered for 90 seconds with a standard high frequency generator, followed by a 1 minute resting period.
  ERCP with SEMS alone (standard of care)
Period: Overall Study
Arm/Group | ERCP With SEMS Plus Radiofrequency Ablation | ERCP With SEMS Alone (Standard of Care)
Started | 13 | 11
Completed | 13 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ERCP With SEMS Plus Radiofrequency Ablation | ERCP With SEMS Alone (Standard of Care) | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Continuous [Mean (Full Range); unit: years] | 62.5 [42 to 84] | 57.9 [44 to 69] | 60.4 [42 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 8 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 11 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 11 | 9 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 11 | 24

OUTCOME MEASURES:

1. Primary Outcome: Rate of Failure
Time Frame: 180 days
Population: Data were not collected
Arm/Group | ERCP With SEMS Plus Radiofrequency Ablation | ERCP With SEMS Alone (Standard of Care)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Rate of Stent Patency
Time Frame: 1 and 3 months post procedure
Population: Data were not collected
Arm/Group | ERCP With SEMS Plus Radiofrequency Ablation | ERCP With SEMS Alone (Standard of Care)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Incidence of Procedure Related Complications
Time Frame: 1 month
Population: Data were not collected
Arm/Group | ERCP With SEMS Plus Radiofrequency Ablation | ERCP With SEMS Alone (Standard of Care)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 180 days
Arm/Group | ERCP With SEMS Plus Radiofrequency Ablation | ERCP With SEMS Alone (Standard of Care)
All-Cause Mortality (participants affected / at risk) | 12/13 | 11/11
Serious Adverse Events (participants affected / at risk) | 4/13 | 4/11
Other Adverse Events (participants affected / at risk) | 13/13 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ERCP With SEMS Plus Radiofrequency Ablation (N=13) | ERCP With SEMS Alone (Standard of Care) (N=11)
Neoplasms ben/mal/unk (inc cyst/polyp) Other, spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 1
Duodenal hemorrhage (Gastrointestinal disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ERCP With SEMS Plus Radiofrequency Ablation (N=13) | ERCP With SEMS Alone (Standard of Care) (N=11)
Anemia (Blood and lymphatic system disorders) | 13 | 11
Hypokalemia (Metabolism and nutrition disorders) | 10 | 7
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 13 | 10
Hypoglycemia (Metabolism and nutrition disorders) | 9 | 5
Hyponatremia (Metabolism and nutrition disorders) | 9 | 7
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 13 | 11
Hypernatremia (Metabolism and nutrition disorders) | 4 | 3
INR increased (Investigations) | 12 | 9
Hypomagnesemia (Metabolism and nutrition disorders) | 7 | 8
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 13 | 11
Hypophosphatemia (Metabolism and nutrition disorders) | 7 | 7
Lipase increased (Investigations) | 2 | 3
Creatinine increased (Investigations) | 5 | 1
Serum amylase increased (Investigations) | 3 | 1
Platelet count decreased (Investigations) | 11 | 7
Blood bilirubin increased (Investigations) | 10 | 11
Lymphocyte count decreased (Investigations) | 7 | 7
Neutrophil count decreased (Investigations) | 6 | 3
White blood cell decreased (Investigations) | 9 | 6
Alkaline phosphatase increased (Investigations) | 11 | 11
Alanine aminotransferase increased (Investigations) | 11 | 10
Aspartate aminotransferase increased (Investigations) | 12 | 11
Activated partial thromboplastin time prolonged (Investigations) | 9 | 5
Fibrinogen decreased (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT02340728/Prot_SAP_000.pdf